CLINICAL TRIAL: NCT00751855
Title: Cortisol Augmentation of Prolonged Exposure Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VISN 3 Mental Illness Research, Education and Clinical Center (U.S. Federal Agency)
Responsible Party: Rachel Yehuda, James J. Peters VA Medical Center
Organization: Bronx VA Medical Center (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YEH-08-044
Record Dates: First submitted 2008-09-11; First posted 2008-09-12 (Estimated); Last update posted 2012-07-27 (Estimated); Status verified 2010-10

CONDITIONS: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Hydrocortisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Prolonged Exposure therapy with Hydrocortisone
  Interventions: Behavioral: Prolonged Exposure therapy; Drug: Hydrocortisone
- 2 (Placebo Comparator): Prolonged Exposure therapy with placebo
  Interventions: Behavioral: Prolonged Exposure therapy; Drug: placebo

INTERVENTIONS:
Behavioral: Prolonged Exposure therapy — 10 weekly sessions
Drug: Hydrocortisone — 30mg 45 minutes prior to each PE session including imaginal exposure (8 total)
  Arms: 1
Drug: placebo — placebo
  Arms: 2

SUMMARY:
This study seeks to examine the efficacy of hydrocortisone administration in the augmentation of the therapeutic effects of Prolonged Exposure (PE) therapy, an empirically tested treatment shown to be effective in the the treatment of posttraumatic stress disorder (PTSD). The augmentation builds on both the translation of neuroscience findings demonstrating the effects of glucocorticoids (GCs) on learning, and on empirical clinical findings from other investigators demonstrating beneficial effects of GCs in reducing traumatic memories in trauma-exposed persons.

ELIGIBILITY:
Inclusion Criteria:

* Veterans who experienced a criterion A trauma while deployed, and a current diagnosis of PTSD with a minimum of 6 months
* Capable of understanding, reading and writing English

Exclusion Criteria:

* Incapable and/or unwilling to provide written informed consent prior to participation
* Unwilling and/or unable to discontinue current psychotherapy
* Regular use of psychotropic medication including antidepressants, benzodiazepines, lithium, mood stabilizers, over-the-counter supplements (melatonin, kava-kava, ephedra)
* Regular use of oral or inhaled steroids
* Significant illness (e.g., type I or II diabetes requiring the use of insulin, HIV, AIDS, seizure disorder, anemia, Lyme disease, etc.)
* The veteran, the veteran's physician, or the study physician think that the veteran's clinical state necessitates the prompt initiation of pharmacotherapy or other treatment that would preclude involvement in the study
* Morbid obesity (VMI > 40)
* Clinically significant laboratory abnormalities as determine during medical clearance procedures
* For women, a positive pregnancy test
* Heavy smoking (more than 2 packs a day)
* Substance and/or alcohol abuse and/or dependence within the previous 6 months
* Response of 3 or 4 on the suicidality items of the HDRS or an assessed serious suicide risk
* Current psychosocial problems that might interfere with treatment compliance
* A lifetime history of schizophrenia, schizoaffective disorder, bipolar disorder, obsessive compulsive disorder or PTSD due to a trauma not sustained in the combat theater

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2008-07; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Change in PTSD symptom severity as assessed by the Clinician Administered PTSD Scale (CAPS) | Baseline (Week 0), endpoint (week 11)

SECONDARY OUTCOMES:
Cognitive performance (learning and retention in an episodic memory task, attention and working memory) | Baseline (Week 0), endpoint (week 11)
Other measures of clinical outcome, psychological state and functioning | Approximately 1 week prior to starting therapy (Week 0) and approximately 1 week after completing 10 weeks of therapy (week 11)
Biological measures associated with PTSD severity | Approximately 1 week prior to starting therapy (Week 0) and approximately 1 week after completing 10 weeks of therapy (week 11)

CONTACTS AND LOCATIONS:
Locations (1):
- James J. Peters Veterans Affairs Medical Center, The Bronx, New York, United States